CLINICAL TRIAL: NCT05637983
Title: Ultrasound-guided Femoral Puncture to Reduce Access- Related Complications After TAVR: (ACCESS-TAVR SIRIO)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Toscana Gabriele Monasterio (Other)
Collaborators: Nicolaus Copernicus University (Other)
Responsible Party: Principal Investigator, Sergio Berti, Director Cardiac Diagnostic and Interventional Unit, Fondazione Toscana Gabriele Monasterio
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Versione: 1.0 del 18/06/2020
Record Dates: First submitted 2022-11-25; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Intervention Model Description: 1:1 randomized trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- US-guided femoral puncture (Experimental): US-guided femoral puncture and Perclose ProGlide/Prostyle implantation during transcatheter aortic valve replacement (TAVR)
  Interventions: Procedure: US-guided femoral puncture vs Fluoroscopy-guided puncture
- Fluoroscopy-guided puncture (Active Comparator): Fluoroscopy-guided puncture and Perclose ProGlide/Prostyle implantation during transcatheter aortic valve replacement (TAVR)
  Interventions: Procedure: US-guided femoral puncture vs Fluoroscopy-guided puncture

INTERVENTIONS:
Procedure: US-guided femoral puncture vs Fluoroscopy-guided puncture — US-guided femoral puncture and Perclose ProGlide®/Prostyle implantation compared to Fluoroscopy-guided puncture and Perclose ProGlide®/Prostyle in TAVR

SUMMARY:
Recent observational data showed a marked reduction of vascular and bleeding complications by the use of ultrasound(US)-guided femoral artery puncture to gain the vascular access and guide the implantation of the Perclose ProGlide® vascular closure system.

We aimed to compare in a 1:1 randomized fashion the effect of US-guided femoral puncture and Perclose ProGlide® implantation optimization vs fluoroscopy-guided puncture followed by Perclose ProGlide/ ProStyle implantation (standard approach) during TAVR.

DETAILED DESCRIPTION:
Transfemoral approach has become the standard route for a transcatheter aortic valve replacement (TAVR) procedure. Despite the technology improvements, vascular complications and access-related bleeding are frequently observed after TAVR and emerge predominantly within 30 days after TAVR. Recent observational data showed a marked reduction of vascular and bleeding complications by the use of ultrasound(US)- guided femoral artery puncture to gain the vascular access and guide the implantation of the Perclose ProGlide® vascular closure system.

We aimed to compare in a 1:1 randomized fashion the effect of US-guided femoral puncture and Perclose ProGlide® implantation optimization vs fluoroscopy-guided puncture followed by Perclose ProGlide/ ProStyle implantation (standard approach) during TAVR.

ELIGIBILITY:
Inclusion Criteria:

* Eligible Patients are male or female with severe aortic stenosis evaluated by the Heart Team as candidate to TAVR based on the current cardiology guidelines.

Exclusion Criteria:

* Refusal to participate in the study;
* Inability to provide written consent to the study protocol;
* Chronic immuno-suppressant therapy;
* Any concomitant condition which, in the opinion of the Investigator, would not allow safe participation in the study (e.g., drug addiction, alcohol abuse, emotional/psychological disorder);
* Enrolment in another study that could confound the results of this study;
* Life expectancy < 1 year;
* Any contraindication to TAVR procedure;
* Non transfemoral TAVR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Estimated)
Dates: Start 2022-07-04 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Composite of CV mortality, vascular complications or access-related bleeding after TAVR at 30 days. | 1 month

SECONDARY OUTCOMES:
CV mortality | 1 month
Vascular complications | 1 month
Life-threatening or disabling bleeding | 1 month
  Fatal bleeding (BARC type 5) OR Bleeding in a critical organ, such as intracranial, intraspinal, intraocular, or pericardial necessitating pericardiocentesis, or intramuscular with compartment syndrome (BARC type 3b and 3c) or Bleeding causing hypovolemic shock or severe hypotension requiring vasopressors or surgery (BARC type 3b) OR Overt source of bleeding with drop in haemoglobin ≥5 g/dl or whole blood or packed red blood cells (RBCs) transfusion ≥4 units (BARC type 3b)
Major bleeding (BARC type 3a) | 1 month
  Overt bleeding either associated with a drop in the haemoglobin level of at least 3.0 g/dl or requiring transfusion of two or three units of whole blood/RBC, or causing hospitalization or permanent injury, or requiring surgery AND Does not meet criteria of life-threatening or disabling bleeding
Major vascular complications | 1 month
  Any aortic dissection, aortic rupture, annulus rupture, left ventricle perforation, or new apical aneurysm/pseudo-aneurysm OR Access site or access-related vascular injury (dissection, stenosis, perforation, rupture, arterio-venous fistula, pseudoaneurysm, haematoma, irreversible nerve injury, compartment syndrome, percutaneous closure device failure) leading to death, lifethreatening or major bleeding, visceral ischaemia, or neurological impairment OR Distal embolization (non-cerebral) from a vascular source requiring surgery or resulting in amputation or irreversible end-organ damage OR The use of unplanned endovascular or surgical intervention associated with death, major bleeding, visceral ischaemia or neurological impairment OR Any new ipsilateral lower extremity ischaemia documented by patient symptoms, physical exam, and/or decreased or absent blood flow on lower extremity angiogram OR Surgery for access siterelated nerve injury OR Permanent access site-related nerve injury
Minor vascular complications | 1 month
  Access site or access-related vascular injury (dissection, stenosis, perforation, rupture, arteriovenous fistula, pseudoaneurysms, haematomas, percutaneous closure device failure) not leading to death, life-threatening or major bleeding, visceral ischaemia, or neurological impairment OR Distal embolization treated with embolectomy and/or thrombectomy and not resulting in amputation or irreversible end-organ damage OR Any unplanned endovascularstenting or unplanned surgical intervention not meeting the criteria for a major vascular complication OR Vascular repair or the need for vascular repair (via surgery, ultrasound-guided compression, transcatheter embolization, or stent-graft) OR Percutaneous closure device failure of a closure device to achieve haemostasis at the arteriotomy site leading to alternative treatment (other than manual compression or adjunctive endovascular ballooning).

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Berti, MD, Principal Investigator — Fondazione Toscana Gabriele Monasterio; Eliano Navarese, Principal Investigator — Nicolaus Copernicus University
Locations (1):
- Fondazione Toscana Gabriele Monasterio, Massa, MS, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Strauss SA, Ma GW, Seo C, Siracuse JJ, Madassery S, Truesdell AG, Pereira K, Korngold EC, Kayssi A. Ultrasound-guided versus anatomic landmark-guided percutaneous femoral artery access. Cochrane Database Syst Rev. 2025 Mar 28;3(3):CD014594. doi: 10.1002/14651858.CD014594.pub2. PMID 40152297